CLINICAL TRIAL: NCT04450355
Title: Effects of Continuous Infusion of Intravenous Nefopam on Postoperative Pain and Opioid Consumption After Video Assisted Thoracic Surgery: A Double Blind Randomized Controlled Trial
Brief Title: Effects of Continuous Infusion of Intravenous Nefopam on Postoperative Pain and Opioid Consumption After VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Pharmbio Korea (Unknown)
Responsible Party: Principal Investigator, Hojin Lee, MD, Clinical assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001-036-1092
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Pain
Keywords: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Nefopam; Saline Solution

STUDY DESIGN:
Intervention Model Description: A prospective randomized double-blinded study
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes assessor not involved in this study will investigate the outcomes. The patient will be not informed of the infusion of nefopam by not attaching an identifiable label so that it cannot be distinguished from normal saline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nefopam group (Experimental): At the end of induction, the nefopam group will receive intravenous nefopam 20mg mixed with 50ml of normal saline, and at the end of surgery, this group will receive intravenous nefopam 60mg mixed with 50ml of normal saline at a rate of 2ml/hr.
  Interventions: Drug: Nefopam 80mg/day
- Control group (Placebo Comparator): The control group will receive intravenous normal saline 50ml at the end of induction and receive intravenous normal saline 50ml at a rate of 2ml/hr at the end of surgery.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Nefopam 80mg/day — continuous nefopam infusion
  Arms: Nefopam group
Drug: Normal saline — continuous normal saline infusion
  Arms: Control group

SUMMARY:
This prospective, randomized, double-blinded study is designed to evaluate the postoperative analgesic effect of the continuous infusion of intravenous nefopam in patients undergoing video-assisted thoracic surgery (VATS). We hypothesize that the continuous infusion of intravenous nefopam can significantly reduce postoperative opioid consumption and pain severity in patients with VATS.

DETAILED DESCRIPTION:
Adult patients undergoing elective unilateral VATS segmentectomy or lobectomy are randomly allocated to receive continuous nefopam infusion (n=45) or not (n=45), in addition to a standard postoperative analgesic regimen comprising of IV fentanyl-based patient-controlled analgesia (PCA). At the end of induction, the nefopam group will receive intravenous nefopam 20mg mixed with 50ml of normal saline, and at the end of surgery this group will receive intravenous nefopam 60mg mixed with 50ml of normal saline at a rate of 2ml/hr. The control group will receive intravenous normal saline 50ml at the end of induction and receive intravenous normal saline 50ml at a rate of 2ml/hr.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective unilateral VATS segmentectomy or lobectomy under general anesthesia
* American Society of Anesthesiologists (ASA) physical classification I-II
* Consent to IV-patient controlled analgesia use
* Willingness and ability to sign an informed consent document

Exclusion Criteria:

* Do not understand our study
* Allergies to anesthetic or analgesic medications
* Continuous local anesthetics infiltration for postoperative pain control
* Patients who receive mechanical ventilation more than 2 hours after surgery
* Pregnancy/Breast feeder
* Medical or psychological disease that can affect the treatment response

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Total fentanyl consumption during 24 hours | postoperative 24 hours
  postoperative fentanyl consumption (mcg) via IV patient controlled analgesia

SECONDARY OUTCOMES:
Total fentanyl consumption | postoperative 48 hours
  postoperative fentanyl consumption (mcg) via IV patient controlled analgesia
Postoperative pain score | postoperative 24, 48 hours
  11-pointed NRS pain score at resting/coughing/movement NRS (0-10): 0, "no pain"; 10, "worst pain imaginable"
Postoperative nausea and vomiting | postoperative 24, 48 hours
  Incidence of postoperative nausea and vomiting (%)
chronic postsurgical pain | 3-months after surgery
  Incidence of chronic postsurgical pain (NRS ≥ 3) (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tirault M, Derrode N, Clevenot D, Rolland D, Fletcher D, Debaene B. The effect of nefopam on morphine overconsumption induced by large-dose remifentanil during propofol anesthesia for major abdominal surgery. Anesth Analg. 2006 Jan;102(1):110-7. doi: 10.1213/01.ANE.0000181103.07170.15. PMID 16368814
- [Background] Du Manoir B, Aubrun F, Langlois M, Le Guern ME, Alquier C, Chauvin M, Fletcher D. Randomized prospective study of the analgesic effect of nefopam after orthopaedic surgery. Br J Anaesth. 2003 Dec;91(6):836-41. doi: 10.1093/bja/aeg264. PMID 14633755